CLINICAL TRIAL: NCT03939767
Title: Evaluation of an eXtended and proacTive Dosing regimEn in Treatment-Naïve Patients With Wet Age-related Macular Degeneration (wAMD)
Brief Title: Assessment of Proactive Treatments in Patients With Wet Age-related Macular Degeneration (wAMD) Which Have Never Undergone Treatment of This Particular Disease
Acronym: XTEND
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 20359
Record Dates: First submitted 2019-05-04; First posted 2019-05-07 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Wet Age-related Macular Degeneration
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- wAMD patients: Patients with a diagnosis of wAMD and naïve to any treatment in the study eye will be enrolled after the decision by treating physician for IVT aflibercept therapy according to the local label.
  Interventions: Drug: Aflibercept (Eylea, BAY86-5321)

INTERVENTIONS:
Drug: Aflibercept (Eylea, BAY86-5321) — As prescribed by the treating physician according to the local label. No IVT aflibercept will be provided due to a nature of observational study.

SUMMARY:
In this observational study researchers want to learn more about changes in visual acuity (clarity of vision) with proactive flexible treatments over time in patients suffering from wet age-related macular degeneration (wAMD) after decision to treat with Aflibercept (Eylea) was made. Wet AMD is an eye disease that progressively destroys the macula, the central portion of the retina, impairing central vision.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of wAMD.
* Patients for whom the decision to initiate treatment with IVT aflibercept in a proactive regimen was made as routine clinical practice.
* Treatment-naïve in the study eye (no prior therapy for wAMD).
* Patient age ≥50 years of age.
* Written informed patient consent before the start of data collection (according to the requirements of the local authorities and laws).

Exclusion Criteria:

* Participation in an investigational program with interventions outside of routine clinical practice.
* Patients with contraindications to IVT aflibercept listed in the local marketing authorization.
* Planned treatment regimen outside of the local marketing authorization.
* Patients with eye diseases, e.g. advanced glaucoma or visually significant cataracts, likely to require surgery during the observation period in the study eye.
* Concomitant ocular or systemic administration of drugs up to 3 months before IVT aflibercept treatment that could interfere with or potentiate the mechanism of action of IVT aflibercept, including other anti-VEGF agents in the fellow eye.
* Any other retinal disease which may interfere with the treatment of wAMD.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 2.000 patients from sites in Asia-Pacific, Europe, Latin America and North America.
Sampling Method: Probability Sample
Enrollment: 1563 (Actual)
Dates: Start 2019-05-12 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-10-17 (Actual)

PRIMARY OUTCOMES:
The change in BCVA (best corrected visual acuity) | Baseline to 12 months
  In treatment-naïve wAMD patients treated with IVT aflibercept in a flexible proactive treatment pattern (fixed dosing or T&E (Treat and Extend Regimen)) by label regimen.

SECONDARY OUTCOMES:
The change in BCVA | Baseline to 24 and 36 months
The change in BCVA by intended treatment regimen | Baseline to 12, 24 and 36 months
The proportion of patients (eyes) gaining or losing a visual acuity compared to baseline | Baseline at 12, 24 and 36 months
  With letter score of ≥ 0 letters, ≥5 letters, ≥ 10 letters, ≥ 15 letters.
The proportion of patients (eyes) achieving a Snellen equivalent of 20/40 or better (approximately 73 ETDRS letters) | At 12, 24 and 36 months
The changes in central retinal thickness (CRT) | Baseline to 12, 24 and 36 months
The number of injections | Baseline to 12, 24 and 36 months
The distribution of the intervals between injections | Up to 36 months

CONTACTS AND LOCATIONS:
Locations (17):
- Many Locations, Multiple Locations, Argentina
- Many Locations, Multiple Locations, Australia
- Many Locations, Multiple Locations, Belgium
- Many Locations, Multiple Locations, Canada
- Many Locations, Multiple Locations, China
- Many Locations, Multiple Locations, Colombia
- Many Locations, Multiple Locations, Denmark
- Many Locations, Multiple Locations, France
- Many Locations, Multiple Locations, Ireland
- Many Locations, Multiple Locations, Italy
- Many Locations, Multiple Locations, Norway
- Many Locations, Multiple Locations, South Korea
- Many Locations, Multiple Locations, Spain
- Many Locations, Multiple Locations, Sweden
- Many Locations, Multiple Locations, Switzerland
- Many Locations, Multiple Locations, Thailand
- Many Locations, Multiple Locations, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- [Derived] Bailey C, Chandran M, Gale R, Narendran N, Talks J, McGoey H, Keshk Z, Morgan-Warren P, Allmeier H, Machewitz T, Patel PJ, Varma D. 2-year results from an observational study of proactive treatment regimens with intravitreal aflibercept 2 mg in patients with nAMD in clinical practice: XTEND study UK cohort. Eye (Lond). 2025 Apr;39(6):1138-1145. doi: 10.1038/s41433-024-03550-y. Epub 2024 Dec 24. PMID 39719502
- [Derived] Korobelnik JF, Chaudhary V, Mitchell P, Kang SW, Tadayoni R, Allmeier H, Lee J, Zhang X, Machewitz T, Bailey C. XTEND: Two-Year Results from a Global Observational Study Investigating Proactive Dosing of Intravitreal Aflibercept in Neovascular Age-Related Macular Degeneration. Ophthalmol Ther. 2024 Mar;13(3):725-738. doi: 10.1007/s40123-023-00867-x. Epub 2024 Jan 10. PMID 38198053
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards — https://clinicaltrials.bayer.com/study/20359